CLINICAL TRIAL: NCT05511506
Title: Comparison Between Cytokines During First and Second Eye Surgeries in Patients With Bilateral Femtosecond Laser-assisted Cataract Surgery
Brief Title: Cytokines in Femtosecond Laser-assisted Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2022-0473
Record Dates: First submitted 2022-08-11; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-01

CONDITIONS: Cataract
Keywords: cataract; cytokine; pain; miosis
MeSH Terms: conditions — Cataract; Pain; Miosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first-eye group (Other)
  Interventions: Other: aqueous humor collection
- second-eye group (Other)
  Interventions: Other: aqueous humor collection

INTERVENTIONS:
Other: aqueous humor collection — Once the laser procedures were finished, the patient was transported to another surgery operating bed. Before the eyeball was opened, 100-200 μL of aqueous humor was obtained from the anterior chamber via an ultra-thin needle through the paracentesis site of cornea.

SUMMARY:
The investigators performed the current study to compare: 1) the pain scores by Visual Analogue Scale; 2) the cytokines concentrations in aqueous humor by human cytokine antibody array; 3) the prostaglandin E2 (PGE2) concentrations by enzyme linked immunosorbent assay (ELISA); 4) the pupil behaviors by Image J between first-eye and second-eye in bilateral cataract patients undergoing sequential femtosecond laser-assisted cataract surgery (FLACS). To our knowledge, this is the first intraindividual study investigating contralateral effect in FLACS. The findings from the current study may broaden our understanding on the mechanism of sympathetic reaction, help to improve clinical performances, and provide strong clinical guidance for cataract surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive cataract patients aged 40-80 years, regardless of gender, with bilateral similar grades of lens opacity, and scheduled for sequential FLACS were enrolled in this study.

Exclusion Criteria:

* history of ocular or systematic inflammatory diseases like uveitis, rheumatism or other autoimmune diseases;
* previous ocular surgery or trauma;
* preoperative glaucoma, zonular weakness, lens dislocation, or poor pupil dilation (measured pupil diameter <5.0 mm) or synechiae;
* use of systemic or topical steroids, non-steroidal anti-inflammatory drugs (NSAIDs), alpha-adrenergic antagonist, or pain relief medications within 1 month prior to surgery;
* patients with baseline eye pain, having anxiety, muscle spasm around the eye or involuntary eye movement disorders which may influence the pain score;
* eyes needing for any other type of anesthesia, failed to obtain > 100 μl aqueous humor (AH) or encountered intra-operative complications like posterior capsule rupture

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
pain scores | through study completion, an average of 1 year
  pain scores of of eyes undergoing sequential FLACS by Visual Analogue Scale (VAS) scoring system, presenting as a numbered line ranging from 0 (no pain) to 10 (unbearable pain) for the severity of ever experienced pain was used. Higher scores mean a worse outcome.
cytokines concentrations | through study completion, an average of 1 year
  Aqueous PGE2 concentrations were determined by using a commercially available Prostaglandin E2 Parameter ELISA Kit (USA R&D Systems, Inc) in accordance with the manufacturer's protocol. Concentrations of 6 selected cytokines (interleukins (IL-1β, IL-1ra, IL-6, IL-8), monocyte chemotactic protein(MCP-1), tumor necrosis factor-α (TNF-α) in aqueous humor were simultaneously measured using Human Luminex Discovery Assay Multiplex Kits (USA R&D Systems, Inc) by using methods that had been previously described.
pupil behaviors | through study completion, an average of 1 year
  the pupil behaviors by Image J between first-eye and second-eye in bilateral cataract patients undergoing sequential FLACS

CONTACTS AND LOCATIONS:
Overall Officials: yu yinhui, MD, Principal Investigator — Second Affiliated Hospital, Medical College of Zhejiang University, Hangzhou, China
Locations (1):
- Second Affiliated Hospital, Medical College of Zhejiang University, Hangzhou, China, Hangzhou, China